CLINICAL TRIAL: NCT04685369
Title: Effectiveness of Anti-VEGF Treatments in Wet AMD in Active Smokers
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Laurence Postelmans, Head of ophtalmology department, Brugmann University Hospital
Other Study IDs: CHUB-Caspers
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active smokers with wet AMD
  Interventions: Other: Medical Data extraction

INTERVENTIONS:
Other: Medical Data extraction — Medical Data extraction

SUMMARY:
" Wet Age-related Macular Degeneration (wet AMD)" is characterized by the appearance of new choroidal vessels. Several clinical studies have shown the effectiveness of intra-vitreous injections of anti-VEGF (bevacizumab, ranibizumab and aflibercept) against these choroidal neovessels. However, some eyes appear to respond less well or be resistant to anti-VEGF injections, which affects visual acuity. To improve the clinical management of patients with wet AMD, it is important to be able to determine which factors determine the response to anti-VEGF treatment.

Non-modifiable factors such as visual acuity or the patient's age at the time of the first injections, the type and size of choroidal neovascularization, as well as certain genetic polymorphisms are known. Two studies, one carried out in Korean patients, the other in different centers in Singapore, New Zealand, Australia and Switzerland showed that active smoking was associated with a poorer response to intra-vitreous injections of ranibizumab, since smoking is also an already well-known modifiable risk factor for the onset of AMD. Another study in the Netherlands shows a poorer visual prognosis after five years of injection treatment in patients who smoke.

This study aims to study the effect of active smoking on the visual prognosis of patients with exudative AMD and treated with anti-VEGF injections in a Belgian cohort.

ELIGIBILITY:
Inclusion Criteria:

* CHU Brugmann Hospital patients
* Patients who received three intra-vitreous injections of ranibizumab, aflibercept or bevacizumab 4 weeks apart as the first intra-vitreous treatment between January 2016 and December 2020.
* Visual acuity measured before the start of the injections (maximum 1 month) and after the series of three injections (4 to 8 weeks after the last injection)
* Patients whose smoking status is known and for whom the following history appears: hypertension, diabetes, taking anti-coagulants or anti-aggregants.

Exclusion Criteria:

* Patients who have already received another intravitreal treatment in the past.
* Patients who have been treated with dynamic phototherapy before or at the same time as the injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the CHU Brugmann Hospital with Wet AMD having received intra-vitreous injections of anti-VEGF, with a known smoking status.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Monoyer chart result | Baseline
  Best corrected visual acuity using a monoyer chart - data collected on one eye only. Monoyer charts are planks with letters displayed: the letters in each row are the same size and the size increases as you go down.
Monoyer chart result | 4 months after baseline
  Best corrected visual acuity using a monoyer chart - data collected on one eye only. Monoyer charts are planks with letters displayed: the letters in each row are the same size and the size increases as you go down.

SECONDARY OUTCOMES:
Central macular thickness | Baseline
  Central macular thickness measured by optical coherence tomography at baseline examination
Central macular thickness | 4 months after baseline
  Central macular thickness measured by optical coherence tomography at final examination
Pigment epithelial detachment | Baseline
  Morphological analysis of the retinal pigment epithelium on optical coherence tomography (OCT), to assess presence or absence of detachment at baseline visit.
Sub-retinal fluid | Baseline
  Morphological analysis of retinal layers on optical coherence tomography (OCT), to assess presence or absence of sub-retinal fluid at baseline visit.
Choroidal neovascularization subtype | Baseline
  Morphological analysis of fluorescein angiography, to assess the type of choroidal neovascularization at baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Caspers, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No